CLINICAL TRIAL: NCT05069415
Title: Visual Performance and Patient Satisfaction With A New Monofocal Intraocular Lens
Brief Title: Monofocal IOL Visual Outcomes When Targeting Mini Monovision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carolina Eyecare Physicians, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CEP 21-001
Record Dates: First submitted 2021-09-13; First posted 2021-10-06 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-01

CONDITIONS: Cataract; Presbyopia
MeSH Terms: conditions — Cataract; Presbyopia

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Emmetropia (Active Comparator): The target refraction for both eyes will be emmetropia (± 0.25 D).
  Interventions: Device: Eyhance IOL
- Mini monovision (Experimental): The target refraction for the dominant eye will be plano (± 0.25 D) and for the non-dominant eye between -0.75D ±0.15.
  Interventions: Device: Eyhance IOL

INTERVENTIONS:
Device: Eyhance IOL — Intraocular lens replaces the natural lens removed during cataract surgery in both eyes. Target emmetropia OU.
Device: Eyhance IOL — Intraocular lens replaces the natural lens removed during cataract surgery in both eyes. Target mini monovision in the non-dominant eye.

SUMMARY:
This study is a 3-month, prospective, up to 2 center, bilateral, randomized subject masked clinical evaluation of a monofocal intraocular lens (IOL) when both eyes are targeted for emmetropia and when the non-dominant eye is targeted for mini monovision (-0.75 D) in patients with or without astigmatism undergoing routine cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is undergoing bilateral cataract extraction with intraocular lens implantation.
* Willing and able to provide written informed consent for participation in the study
* Willing and able to comply with scheduled visits and other study procedures.
* Scheduled to undergo standard cataract surgery in both eyes within 6 - 30 days between surgeries.
* Subjects who require an IOL power in the range of +5.0 D to +34.0 D only.
* Potential postoperative visual acuity of 0.2 logMAR (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

* Severe preoperative ocular pathology: amblyopia, rubella cataract, proliferative diabetic retinopathy, shallow anterior chamber, macular edema, retinal detachment, aniridia or iris atrophy, uveitis, history of iritis, iris neovascularization, medically uncontrolled glaucoma, microphthalmos or macrophthalmos, optic nerve atrophy, macular degeneration (with anticipated best postoperative visual acuity less than 20/30), advanced glaucomatous damage, etc.
* Uncontrolled diabetes.
* Use of any systemic or topical drug known to interfere with visual performance.
* Contact lens use during the active treatment portion of the trial.
* Any concurrent infectious/non-infectious conjunctivitis, keratitis or uveitis.
* Clinically significant corneal dystrophy.
* Irregular astigmatism.
* History of chronic intraocular inflammation.
* History of retinal detachment.
* Pseudoexfoliation syndrome or any other condition that has the potential to weaken the zonules.
* Previous intraocular surgery.
* Previous refractive surgery.
* Previous keratoplasty
* Severe dry eye
* Pupil abnormalities
* Subject who may reasonably be expected to require a secondary surgical intervention at any time during the study (other than YAG capsulotomy, i.e. LASIK)
* Anesthesia other than topical anesthesia (i.e. retrobulbar, general, etc).
* Any clinically significant, serious or severe medical or psychiatric condition that may increase the risk associated with study participation or may interfere with the interpretation of study results.
* Participation in (or current participation) any ophthalmic investigational drug or ophthalmic device trial within the previous 30 days prior to the start date of this trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry D Solomon, Principal Investigator — Carolina Eyecare Physicians
Locations (2):
- United States (2):
  - Center for Sight, Sarasota, Florida
  - Carolina Eyecare Physicians, LLC, Mt. Pleasant, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Emmetropia | Mini Monovision
Started | 38 | 37
Completed | 34 | 37
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Emmetropia | Mini Monovision | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.1 (6.1) | 69.5 (4.3) | 69.8 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 44
  Male | 13 | 14 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 8 | 13
  White | 29 | 29 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Binocular Distance-corrected Intermediate (66 cm) Visual Acuity at 3 Months.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Emmetropia | Mini Monovision
Number analyzed (Participants) | 34 | 37
logMAR | 0.19 (0.16) | 0.04 (0.10)

2. Secondary Outcome: Binocular Low Contrast Distance Visual Acuity at 3 Months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Emmetropia | Mini Monovision
Number analyzed (Participants) | 34 | 37
logMAR | 0.15 (0.09) | 0.15 (0.13)

3. Secondary Outcome: Distance-corrected Near Visual Acuity at Best Distance at 3 Months
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Emmetropia | Mini Monovision
Number analyzed (Participants) | 34 | 37
logMAR | 0.43 (0.18) | 0.21 (0.15)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Emmetropia | Mini Monovision
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/37
Serious Adverse Events (participants affected / at risk) | 2/34 | 0/37
Other Adverse Events (participants affected / at risk) | 0/34 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Emmetropia (N=34) | Mini Monovision (N=37)
Central retinal vein occlusion (Eye disorders) | 1 | 0
Ischemic optic neuropathy (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/15/NCT05069415/Prot_SAP_000.pdf